CLINICAL TRIAL: NCT02370368
Title: A Comparison of a Dance Programme Delivered With the XBOX Kinect With Traditional Agility Ladder Drills on Agility Scores of Club Level Volleyball Players of the University of the West Indies, Mona
Brief Title: Comparison of Videogame Based Dance Training With Agility Ladder Drills on Agility of Volleyball Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of The West Indies (Other)
Responsible Party: Principal Investigator, Sharmella Roopchand-Martin, Lecturer, The University of The West Indies
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ECP213-13-14
Record Dates: First submitted 2015-02-17; First posted 2015-02-24 (Estimated); Results first posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Healthy Athletes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dance Group (Experimental): Training: participants will engage in dance training with the Xbox Kinect 360 using the Just Dance 2014 disc.
  Duration : 45 minutes per session. Frequency: three times per week for six weeks.
  Interventions: Device: XBOX Kinect Just Dance 2014
- Ladder Drills (Active Comparator): Intervention: Agility ladder drill training. Duration: 45 minutes per session. Frequency: three times per week for six weeks
  Interventions: Other: Agility Ladder Drills

INTERVENTIONS:
Device: XBOX Kinect Just Dance 2014 — The XBOX Kinect Just dance 2014 is videogame based interactive dance programme designed to encourage activity while gaming.
  Arms: Dance Group
Other: Agility Ladder Drills — Types of ladder drill exercises including single leg hop right and left leg, bunny hop, slalom jumps, bunny twist, lateral runs right and left, high knees with forward progression, backward run, bunny hop backward, single leg lateral hops, lateral bunny hops and snake carrioca moguls.
  Arms: Ladder Drills

SUMMARY:
This study will examine the effects of six week dance training, using the Xbox Kinect Just Dance 2014 programme, on the agility scores along with general and hamstring flexibility and extensibility of the hip flexor. The effects of the dance programme will be compared with those of proven agility training techniques (ladder drills).

DETAILED DESCRIPTION:
A randomised clinical trial will be used consisting of 34 (17 in each group) athletes undergoing training. Both groups will undergo one hour of training three times weekly for six weeks, with one group doing dance training (DT) using the Xbox Kinect and the other doing standard training (ST) using traditional ladder drills. Outcomes will be assessed using the Illinois Agility test for agility, sit and reach test for general flexibility, straight leg raise test for hamstring flexibility and the Thomas test for hip flexor extensibility.

ELIGIBILITY:
Inclusion Criteria:

* To be included in the study persons must be playing volleyball at the University of the West Indies at competitive levels and will be required to give written consent to participate in the study.

Exclusion Criteria:

- 1. Anyone who currently has a musculoskeletal injury of the lower limb that prevents them from performing the respective activities.

2. Anyone involved in a dance programme as this will confound the results of the study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2014-09; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
Submit article to a sports journal. Presentation of findings to the athletes and their team captain.

RESULTS

PARTICIPANT FLOW:
Groups:
- Dance Training: Participated in dance training with the XBOX Kinect 3 days per week for six weeks.
- Ladder Drills: Participated in a ladder drill training programme three times per week for six weeks.
Period: Overall Study
Arm/Group | Dance Training | Ladder Drills
Started | 14 | 13
Completed | 8 | 7
Not Completed | 6 | 6
Not completed — Adverse Event | 1 | 2
Not completed — Withdrawal by Subject | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Dance Training: Dance training with the XBOX Kinect 3 times per week for six weeks.
- Ladder Drills: Agility ladder drills 3 times per week for six weeks
- Total: Total of all reporting groups
Arm/Group | Dance Training | Ladder Drills | Total
Number analyzed (Participants) | 14 | 13 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.36 (5.66) | 23.54 (5.27) | 23.96 (5.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 5 | 7 | 12
Region of Enrollment [Number; unit: participants] — All volleyball players currently playing competitively for The University of the West Indies, Jamaica who met the inclusion criteria were recruited for the study.
  participants
    Jamaica | 14 | 13 | 27

OUTCOME MEASURES:

1. Primary Outcome: Change in Agility From Baseline to 6 Weeks
Description: Illinois Agility Test - The athlete is timed during completion of a marked out course
Time Frame: baseline and at 6 weeks
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Dance Training | Ladder Drills
Number analyzed (Participants) | 8 | 7
Seconds | 1.56 (0.5) | 0.86 (0.5)

2. Secondary Outcome: Change in Hamstring Extensibility From Baseline to 6 Weeks
Description: Straight leg raise test - the person lies on their back and are asked to lift the leg straight up trying to keep the knee straight. The knee angle is measured with a goniometer.
Time Frame: Baseline and at 6 weeks
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Dance Training | Ladder Drills
Number analyzed (Participants) | 8 | 7
degrees | 14.6 (13.29) | 7.43 (11.26)

3. Secondary Outcome: Change in Hip Flexor Extensibility From Baseline to 6 Weeks
Description: Thomas test - person lies on their back with the one leg held close to the chest and the other hanging off the bed. The angle at the knee is measured with a goniometer.
Time Frame: baseline and at 6 weeks
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Dance Training | Ladder Drills
Number analyzed (Participants) | 8 | 7
degrees | 21.87 (13.46) | 8.57 (17.38)

ADVERSE EVENTS:
Time Frame: Data on adverse events was collected for the duration of the study which ran from September 2014 to January 2015. Persons were assessed at the beginning and end of every training session for the entire duration of the study's intervention, approximately six weeks per participant. Participants were advised that they could report any adverse events at any point during the research process.
Description: At the beginning and end of every training session participants were asked to indicate if they had any aches, pains or injuries. They were asked to indicate all problems even if they did not think it was related to the training programme.
Arm/Group | Dance Training | Ladder Drills
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 1/8 | 2/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dance Training (N=8) | Ladder Drills (N=7)
Minor musculoskeletal strain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) — One person had ankle pain and two had pain and swelling of the knee. All participants discontinued the study and injuries were treated with anti-inflammatory medications and physical therapy.

LIMITATIONS AND CAVEATS:
The total number of athletes who were eligible for the trial were already small and with drop outs and injuries the resulting group for analysis was small.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No